CLINICAL TRIAL: NCT06200506
Title: Efficacy of Radiofrequency in Primary Dysmenorrhea
Acronym: Rdismenorrea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCompluMadrid
Record Dates: First submitted 2023-11-28; First posted 2024-01-11 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-03

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Physical therapy modality; Diathermy
MeSH Terms: conditions — Dysmenorrhea; Fever

STUDY DESIGN:
Intervention Model Description: Study of a prospective longitudinal clinical trial: two intervention groups and a control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transabdominal radiofrequency application (Experimental): Tecartherapy equipment (Capenergy CM500) specially designed for Uro-Gynecological Physiotherapy will be used.
  A transabdominal radiofrequency application will be performed, with a suprapubic active plate and a passive plate at the sacral level.
  Patient position: Supine position. Sessions:9 Duration: 20 minutes Total intervention: 3 weeks Frequency: 3 times a week sessions will be held three times a week for three weeks
  Interventions: Device: Transabdominal radiofrecuency application
- Intracavitary radiofrequency application (Experimental): Tecartherapy equipment (Capenergy CM500) specially designed for Uro-Gynecological Physiotherapy will be used.
  An intracavitary vaginal radiofrequency application will be performed, with an active intracavitary head and with a fixed plate at the sacral level.
  Patient position: Supine position. Sessions:9 Duration: 20 minutes Total intervention: 3 weeks Frequency: 3 times a week sessions will be held three times a week for three weeks
  Interventions: Device: Intracavitary radiofrequency application
- Control Group (No Intervention): Not treatment received

INTERVENTIONS:
Device: Transabdominal radiofrecuency application — A transabdominal radiofrequency application will be performed, with a suprapubic active plate and a passive plate at the sacral level.
  Patient position: Supine position. Sessions:9 Duration: 20 minutes Total intervention: 3 weeks.
  Frequency: 3 times a week sessions will be held three times a week for three weeks
  Arms: Transabdominal radiofrequency application
Device: Intracavitary radiofrequency application — An intracavitary vaginal radiofrequency application will be performed, with an active intracavitary head and with a fixed plate at the sacral level.
  Patient position: Supine position. Sessions:9 Duration: 20 minutes Total intervention: 3 weeks. Frequency: 3 times a week sessions will be held three times a week for three weeks.
  Arms: Intracavitary radiofrequency application

SUMMARY:
The main objective of the study is to evaluate the effect of radiofrequency on pain associated with primary dysmenorrhea.

The data collected will be: Intensity of pain with the Numeric Pain Rating Scale (NPRS), pressure pain at three points of referred pain from the gynecological system, need or not to take medication, general quality of life with the SF-12 (short form 12) and quality of life in relation to menstruation with the CVM-22. They will be collected at the start of treatment, after the first post-intervention menstruation and after the second post-intervention menstruation.

This study is a randomized clinical trial with two intervention groups and a control group, whose study population is women with primary dysmenorrhea.

The sample size has been calculated with the G* Power 1.9.7 software using repeated measures ANOVA, assuming a two-sided significance level (α=0.05) and 90% power (β=0.10) and 10% losses. A sample of 45 participants (n) was determined to detect a significant change of 1.5 points in the variable measured with the NRS. Forty-five participants were included in this study. In the two intervention groups, radiofrequency will be applied (20 minute sessions for 3 weeks with a frequency of 3 times/week), transabdominal in one group and intravaginal in the other.

Participants must be women between 18 and 35 years old, with regular menstrual cycles (22-38 days according to FIGO), be nulliparous and also not present any of the exclusion criteria detailed in the study.

The data obtained will be analyzed and compared between the different groups in order to draw conclusions.

DETAILED DESCRIPTION:
Dysmenorrhea is a gynecological clinical entity that can be defined as menstrual pain. It usually begins a couple of days before the bleeding or coinciding with the start of the bleeding and usually lasts between 8 and 72 hours.

The main symptom is pelvic and / or abdominal pain that can spread to the lower back or lower limbs. On a psychological level, it associates pictures of depression, anxiety or irritability. It also affects in a very negative way the quality of life, work and / or academic performance (causing episodes of absenteeism) and the social sphere of the women who suffer from it.

In recent years, alternative treatments to pharmacological treatments have been gaining strength, among which physiotherapy stands out. Techniques such as manual therapy, transcutaneous electrical nerve stimulation (TENS), thermotherapy, kinesiology tape, stretching, therapeutic exercises ... are applied in women with primary dysmenorrhea and have been evaluated in numerous studies, most of which are of poor methodological quality.

In clinical practice, one of the physiotherapy modalities that has been applied the most in urogynecological pathologies in women is radiofrequency. Radiofrequency is a physiotherapy intervention that consists of the transfer of energy to the tissues in a resistive or capacitive way using wave frequencies between 0.5 and 1.5 megahertz (MHz). However, at present, there are no clinical trials randomized and controlled that evaluates the effectiveness of radiofrequency in any urogynecological pathology, including primary dysmenorrhea.

Objective: The aim of this study is to assess the effect of radiofrequency on pain associated with primary dysmenorrhea.

Study Type: Randomized controlled clinical trial with two intervention groups and one control group. In the two intervention groups, radiofrequency will be applied (20-minute sessions for 3 weeks with a frequency of 3 times / week). In one of the two groups the application of radiofrequency will be intracavitary and in the other group it will be transabdominal. The control group will not receive any intervention, with the commitment to treat once the study is finished.

Study subjects: Women between 18 and 35 years old, nulliparous, with menstrual pain attributable to primary dysmenorrhea (self-reported pain in most menstrual cycles and at least in the last three menstrual cycles).

Sample size: The sample size was calculated to identify clinically relevant effects on the primary outcome, numerical pain rating scale.

The sample size has been calculated with the G* Power 1.9.7 software using repeated measures ANOVA, assuming a two-sided significance level (α=0.05) and 90% power (β=0.10) and 10% losses. A sample of 45 participants (n) was determined to detect a significant change of 1.5 points in the variable measured with the NRS. Forty-five participants would be required to detect a significant change, 15 in each group.

Interventions:

Intervention group 1 (G1): A transabdominal application (fixed plate at the sacral level) will be performed.

Intervention group 2 (G2): A vaginal intracavitary application (fixed plate at the sacral level) will be performed.

Control group (C): No intervention will be carried out, with the commitment to carry out a postponed intervention in case of having positive results in the study.

Outcomes:

Primary Outcome Measure:

• Numerical Pain Rating Scale.

Secondary Outcome Measures:

* Questionnaire on quality of life in relation to menstruation (CVM-22), validated in Spanish.
* Pressure Pain Threshold (PPT) in the abdominal region recorded in previous studies.
* Number and quantity of analgesics, anti-inflammatories taken to alleviate the pain.

Key words: Dysmenorrhea, physical therapy modality, diathermy, thermotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years.
* Menstrual pain: During bleeding and/or the previous 48 hours.
* Nulliparous.
* Regular menstrual cycles (24-38 days according to FIGO).

Exclusion Criteria:

* Currently using contraceptives that prevent intracavitary application (hormonal intrauterine devices and vaginal rings).
* Have any recent abdominal or pelvic surgery that prevents the application of intra/extracavitary heat.
* Dysmenorrhea secondary to other gynecological pathologies (endometriosis, adenomyosis, uterine fibroids...)
* Pregnancy.
* Have received physiotherapy treatment for the painful episode in the six months prior to the study.
* To present situations of contraindication of diathermy, radiofrequency or tecartherapy: implanted devices that work with batteries (pacemakers), metallic implants near the lumbopelvic region, uncontrolled or recent cancer processes, recent hemorrhages, alterations in sensitivity in the area to be treated , local active infections near the region to be treated, febrile states, skin wounds and epileptic processes.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with menstrual pain
Enrollment: 45 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Dysmenorrheal pain intensity | Baseline
  Dysmenorrheal pain intensity (measured using the NPRS scale) at rest. It will be evaluated three times with 1 minute between the three evaluations and the average will be noted.
Dysmenorrheal pain intensity | One month
  Dysmenorrheal pain intensity (measured using the NPRS scale) at rest. It will be evaluated three times with 1 minute between the three evaluations and the average will be noted.
Dysmenorrheal pain intensity | Two month
  Dysmenorrheal pain intensity (measured using the NPRS scale) at rest. It will be evaluated three times with 1 minute between the three evaluations and the average will be noted.

SECONDARY OUTCOMES:
Quality of life during menstruation. | Baseline
  Quality of life during menstruation, assessed with the previously validated Spanish version of the CVM-22 questionnaire.
Quality of life during menstruation. | One month
  Quality of life during menstruation, assessed with the previously validated Spanish version of the CVM-22 questionnaire.
Quality of life during menstruation. | Two month
  Quality of life during menstruation, assessed with the previously validated Spanish version of the CVM-22 questionnaire.
Quality of life (General) | Baseline
  Quality of life during, assessed with the previously validated Spanish version of the SF-12 questionnaire.
Quality of life (General) | One month
  Quality of life during, assessed with the previously validated Spanish version of the SF-12 questionnaire.
Quality of life (General) | Two month
  Quality of life during, assessed with the previously validated Spanish version of the SF-12 questionnaire.
Pressure Pain Threshold | Baseline
  Painful sensitivity to pressure at three points in the abdominal region (suprapubic, at the oblique minor reference points according to the protocol), recorded with a digital algometer, Jtech Medical Commander algometer.
Pressure Pain Threshold | One month
  Painful sensitivity to pressure at three points in the abdominal region (suprapubic, at the oblique minor reference points according to the protocol), recorded with a digital algometer, Jtech Medical Commander algometer.
Pressure Pain Threshold | Two month
  Painful sensitivity to pressure at three points in the abdominal region (suprapubic, at the oblique minor reference points according to the protocol), recorded with a digital algometer, Jtech Medical Commander algometer.
Number and quantity of drugs. | Baseline
  Consumption of drugs due to the current episode. The patient was asked what drugs he was taking, and the second investigator from the Complutense University of Madrid will classify the dosage as "non-use", "occasional use", "regulated use", "use greater than the prescribed". This same researcher classified each drug according to its action as: analgesics, anti-inflammatories, muscle relaxants, psychoactive drugs (anxiolytics, antidepressants) and other drugs.
Number and quantity of drugs. | One month
  Consumption of drugs due to the current episode. The patient was asked what drugs he was taking, and the second investigator from the Complutense University of Madrid will classify the dosage as "non-use", "occasional use", "regulated use", "use greater than the prescribed". This same researcher classified each drug according to its action as: analgesics, anti-inflammatories, muscle relaxants, psychoactive drugs (anxiolytics, antidepressants) and other drugs.
Number and quantity of drugs. | Two month
  Consumption of drugs due to the current episode. The patient was asked what drugs he was taking, and the second investigator from the Complutense University of Madrid will classify the dosage as "non-use", "occasional use", "regulated use", "use greater than the prescribed". This same researcher classified each drug according to its action as: analgesics, anti-inflammatories, muscle relaxants, psychoactive drugs (anxiolytics, antidepressants) and other drugs.

CONTACTS AND LOCATIONS:
Overall Officials: MARÍA JOSÉ DÍAZ-ARRIBAS, PhD, Study Director — UCM
Locations (1):
- Universidad Complutense de Madrid, Madrid, Madrid, Spain